CLINICAL TRIAL: NCT04391738
Title: Relationship Between Obesity and Severe Acute Respiratory Syndrome Coronavirus-2 in Patient With SARS-CoV-2 Admitted in Intensive Care : A Multicenter Retrospective Cohort Study
Brief Title: Association Between BMI and COVID-19
Acronym: BMI-SARS-CoV-2
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: DEC20-095
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV 2
Keywords: Intensive Care; Invasive Mechanical Ventilation; Body Mass Index; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BMI SARS-CoV-2: Patients admitted to Intensive Care Unit with SARS-CoV-2
  Interventions: Other: Patients admitted to Intensive Care Unit with SARS-CoV2

INTERVENTIONS:
Other: Patients admitted to Intensive Care Unit with SARS-CoV2 — Patients admitted to Intensive Care Unit with SARS-CoV2

SUMMARY:
This study will involve collection of pseudonymized data from hospital-based data reporting at multiple international sites. Collating data from a large volume of patients with COVID-19 admitted in ICU across multiple international sites will enable investigation of whether obesity is a risk factor for complicated from of SARS-CoV-2 in adult patients and whether this association is independent of other cardiometabolic risk factors.

DETAILED DESCRIPTION:
The COVID-19 pandemic is characterized by a high frequency of patients with severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), who often require invasive mechanical ventilation (IMV). Body mass index (BMI) was however rarely mentioned in early clinical reports.

Disease severity gradually increased with body mass index (BMI) categories among patients admitted in intensive care unit (ICU) for severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), the need for invasive mechanical ventilation (IMV), reaching 85% in patients with class II or III obesity ( BMI > 35 kg/m2).

In summary, there is an urgent need for more evidence on the specific role played by obesity in the development of COVID-19 complications, and more particularly of severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2)

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged 18 years or over
* Has been admitted to ICU with COVID-19 disease.
* COVID-19 disease has been confirmed by PCR for SARS-CoV-2
* Height and weight or BMI on admission has been recorded
* Data has been collected in an ethical manner as part of a national database or clinical auditing process approved by the local institution or collaboration

Exclusion Criteria:

-There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to Intensive Care Unit for SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Relationship between body mass index (BMI) and SARS-CoV-2 | 3 months
  The primary objective of this study is to investigate the relationship between obesity, as determined by body mass index (BMI), and severe pneumonia, as defined by the need of invasive mechanical ventilation ( IMV), among patient admitted in ICU for SARS-CoV-2, across multiple centers, in multiple countries.

SECONDARY OUTCOMES:
Associations between BMI and outcomes is independent of the known cardiometabolic risk factors | 3 months
  Investigate whether the associations between BMI and outcomes is independent of the known cardiometabolic risk factors, hypertension, diabetes, dyslipidemia, and current smoking.
Investigate the modifying effects of age and sex on the associations between BMI and outcome: Invasive mechanical ventilation | 3 months
  Investigate the modifying effects of age and sex on the associations between BMI and outcome: Invasive mechanical ventilation
Investigate the modifying effects of age and sex on the associations between BMI and outcome: mortality | 3 months
  Investigate the modifying effects of age and sex on the associations between BMI and outcome: mortality

CONTACTS AND LOCATIONS:
Overall Officials: Francois Pattou, MD, Study Director — Centre Hospitalier Régional & Universitaire de Lille (CHRU)
Locations (1):
- Centre Hospitalier Régional & Universitaire de Lille (CHRU), Lille, France